CLINICAL TRIAL: NCT00657293
Title: Arm Training in COPD: Short and Medium Term Effects on Dyspnoea, Health-related Quality of Life, Arm Function and Arm Exercise Capacity.
Brief Title: Arm Training in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Dr. Roger Goldstein, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Goldstein_Arm1207
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; arm training; dyspnoea; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C (Sham Comparator): In an attempt to make the groups comparable in terms of attention, the control group will receive a sham.
  Interventions: Behavioral: Purdue pegboard test (sham)
- ATP (Active Comparator): Patients will undergo a specific arm training program (ATP).
  Interventions: Behavioral: Arm training program

INTERVENTIONS:
Behavioral: Arm training program — Patients will undergo a specific arm training program (ATP) three times a week for the duration of the 6 week program. The ATP will consist predominantly of resistance exercises. Muscle groups targeted during the ATP will include deltoid, biceps and triceps, pectoralis and latissimus. Subjects will train using multi station gym equipment and free weights.
  Arms: ATP
Behavioral: Purdue pegboard test (sham) — In an attempt to make the groups comparable in terms of attention, the control group will perform the purdue pegboard test of finger dexterity. The tasks will be performed in a sitting position with the arms supported on a table. This test will consist of 4 timed tasks where as many pins as possible will be placed on a pegboard in a given time. Performance of the pegboard test is likely to improve with practice which may serve to motivate the patients to continue practicing over the 6-week period. Subjects will perform this activity 3 times per week with supervision provided by a physiotherapist.
  Arms: C

SUMMARY:
Patients with chronic lung disease often report shortness of breath when they use their arms for simple activities of daily living such as dressing, lifting, shaving, bathing and brushing their hair and teeth. The best type of arm training for these patients is still unknown.

The objectives of this study are to:

* develop a feasible and safe arm training program (ATP) for these patients;
* examine the effects of this ATP on quality of life, arm function, arm exercise capacity and symptoms during activities of daily living;
* examine the effects of ATP on breathing responses during arm exercises.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common condition throughout Canada and the rest of the world. Patients with COPD often describe of breathlessness that makes it difficult for them to participate in physical activity. Specifically, patients often report shortness of breath when they use their arms for simple activities of daily living such as dressing, lifting and bathing. Exercise training has been shown to reduce breathlessness in people with COPD. Compared with studies that have looked at the effects of exercise using the leg muscles, studies that focus on training the arm muscles in people with COPD are sparse. Although earlier work shows that arm training increases arm exercise capacity, the effects on other measures such as breathlessness are not clear. Therefore, the objectives of this study are; (i) to develop a feasible and safe arm training program (ATP) for patients with COPD based on the best available evidence, (ii) to examine the effectiveness of this ATP on breathlessness during activities of daily living, health-related quality of life, arm function and arm exercise capacity, (iii) to examine the physiological mechanisms underpinning any change in these outcomes in response to the ATP.

Patients with COPD will be assigned by chance to either a treatment or control group. All patients in both groups will complete the 6-week pulmonary rehabilitation (PR) program that is well-established at our centre (West Park). During this program all patients will complete leg exercises, such as walking or cycling, and receive education about how to best manage their disease. In addition to this PR program, the treatment group will complete a specific ATP involving overhead arm exercises and free weights. The control group will undergo a "sham" ATP consisting of finger exercises. Before and after the ATP we will collect measures of; (i) breathlessness during activities of daily living, fatigue and quality of life, (ii) arm exercise capacity, (iii) arm function and, (iv) arm muscle force. During the tests of arm exercise capacity a special machine (breathing-gas analysis system) will be worn. Measurements will be compared between the treatment and control groups before, immediately after the ATP and also 3 months after completing the ATP.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD
* a forced expiratory volume in one second (FEV1) of less than 80% the predicted normal value
* must report dyspnoea during at least one activity of daily living that requires arm activity
* must have a smoking history greater than 10 pack years and
* must be able to provide written informed consent

Exclusion Criteria:

* acute exacerbation of COPD that required a change in pharmacological management within the preceding two months
* an inability to understand English
* cognitive impairment
* requirement for mechanical ventilation for all or part of the day
* tapering doses of oral corticosteroids or xanthines
* evidence of a musculoskeletal or neurological condition which could adversely affect arm exercise performance
* symptomatic ischemic cardiac disease
* a history of previous lung surgery and alpha1 antitrypsin deficient emphysema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Feasibility measures, dyspnoea during activities of daily living, fatigue, health-related quality of life, unsupported arm exercise capacity, arm function and peripheral muscle force | Primary outcome measures will be collected before PR program, on completion of the PR program (at 6 weeks) and at three months following completion of the PR program.

SECONDARY OUTCOMES:
Peak cardiorespiratory responses during incremental unsupported upper limb exercise test | Secondary outcome measures will be collected before PR program, on completion of the PR program (at 6 weeks) and at three months following completion of the PR program.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, M.D., Principal Investigator — West Park Healthcare Centre; Dina Brooks, Ph.D., Principal Investigator — West Park Healthcare Centre; Tania Janaudis-Ferreira, Msc, Study Chair — West Park Healthcare Centre; Kylie Hill, Ph.D., Study Chair — West Park Healthcare Centre; Tom Dolmage, Msc, Study Chair — West Park Healthcare Centre; Marla Beauchamp, Msc, Study Chair — West Park Healthcare Centre; Karin Wadell, Ph.D., Study Chair — Umea University
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada